CLINICAL TRIAL: NCT06943690
Title: Safety and Efficacy Study of Single-port Robotic Versus Multi-port Robotic Radical Rectal Cancer Surgery: A Multi-center, Prospective, Open Label, Non-inferiority, Randomized Controlled Trial
Brief Title: Safety and Efficacy Study of Single-port Robotic Versus Multi-port Robotic Radical Rectal Cancer Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shandong Provincial Hospital (Other Government); First Affiliated Hospital of Wenzhou Medical University (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhao Ren, Chief Physicion, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RASILS-01
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Rectal Cancer; Surgery
Keywords: Rectal Cancer; Robotic Surgery
MeSH Terms: conditions — Rectal Neoplasms | interventions — sperm releasing substance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-Port Robotic Surgery (Experimental): Patients with rectal cancer undergo single-port robotic surgery.
  Interventions: Procedure: Single-port robotic surgery
- Multi-Port Robotic Surgery (Active Comparator): Patients with rectal cancer undergo multi-port robotic surgery.
  Interventions: Procedure: Multi-port robotic surgery

INTERVENTIONS:
Procedure: Single-port robotic surgery — In this group, patients will be operated using a single-port surgical robot system. In the single-port configuration, a four-channel trocar shall be used. The surgical tools are steered through the curved access channels in the trocar to enter a patient's abdomen. The surgical procedure followed the principle of total mesorectal excision.
  Other Names: SPRS
  Arms: Single-Port Robotic Surgery
Procedure: Multi-port robotic surgery — In this group, patients will be operated using a multi-port surgical robot system. Surgical instruments enter the abdominal cavity through 4 separate trocars. The surgical procedure followed the principle of total mesorectal excision.
  Other Names: MPRS
  Arms: Multi-Port Robotic Surgery

SUMMARY:
This study is designed to evaluate the safety and efficacy of single-port robotic surgery compared to multi-port robotic surgery for rectal cancer.

DETAILED DESCRIPTION:
Surgical robots were born in the 1980s and have the advantages of being precise, flexible, less invasive and remotely operable than traditional surgical methods. The single-port robot is a further extension of minimally invasive surgery by placing multiple instruments through a single incision. Most studies have reported on the perioperative outcomes of robotic versus conventional laparoscopic surgery in the treatment of colorectal cancer. However, there are limited data comparing the perioperative outcomes of single-port robotics and multi-port robotics in the treatment of colorectal cancer，especially in rectal cancer surgery. The purpose of this study is to evaluate the safety and efficacy of single-port robotic surgery compared to multi-port robotic surgery for rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years < age ≤80 years
* Tumor located in the mid to high rectum (lower edge of tumor ≥ 5 cm from anal verge)
* Pathological rectal carcinoma
* Clinically diagnosed c/ycT1-3N0-1M0 lesions according to the 8th Edition of AJCC Cancer Staging Manual
* Tumor size of 10 cm or less
* No history of other malignant tumors
* ECOG score is 0-1
* ASA score is Ⅰ-Ⅲ
* Informed consent

Exclusion Criteria:

* Body mass index (BMI) >35 kg/m2
* Familial adenomatous polyposis (FAP)
* Inflammatory bowel disease (IBD)
* Multiple malignant colorectal tumors
* Pregnant woman or lactating woman
* Severe mental disease
* Previous gastrointestinal surgery (except appendectomy ）
* Combination of intestinal obstruction, bleeding, perforation requiring emergency surgery
* Requirement of simultaneous surgery for other disease
* Serious disorders of liver and kidney function, coagulation function, or severe underlying diseases that cannot tolerate the surgery.
* Patients or family members who cannot understand the study program.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Surgical success rate | intraoperative
  Proportion of robotic procedures not converted to laparoscopic or open surgery

SECONDARY OUTCOMES:
Operative time | intraoperative
  Operative time（minutes）
Intraoperative blood loss | intraoperative
  Estimated blood loss（milliliters，ml）
Incision length | intraoperative
  Incision length（centimeters，cm）
Total incision length | intraoperative
  The sum of all incision lengths（centimeters，cm）
Length of stay | 1-30 days after surgery
  The postoperative day when patients complied with the predefined discharge
Postoperative recovery course | 1-14 days after surgery
  Time to first ambulation, flatus, liquid diet and semi-liquid diet （hours after surgery）
Early morbidity rate | 30 days after surgery
  morbidity rate 30 days after surgery
Pain score | 1-3 days after surgery
  postoperative pain is recorded using the visual analog scale (VAS) pain score （0-10 points）tool on postoperative day 1, 2, 3
Tumor size | 14 days after surgery
  The diameter of tumors（centimeters，cm）
Incisal margin | 14 days after surgery
  Length of proximal and distal margin （centimeters，cm）
Lymph node detection | 14 days after surgery
  Lymph nodes harvested（numbers）
Cosmetic effect | 1 month, 6 months and 1 year after surgery
  European Organization for Research and Treatment of Cancer Quality of Life
The quality of life-Colorectal | 1 month, 6 months and 1 year after surgery
  European Organization for Research and Treatment of Cancer Quality of Life
disease free survival rate | 12 months after surgery
  1-year disease free survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Ren Zhao, MD, PHD, Principal Investigator — Ruijin Hospitlal , Shanghai Jiaotong University School of Medicine; Leping Li, MD, Study Director — Shandong Provincial Hospital; Xian Shen, MD, Study Director — First Affiliated Hospital of Wenzhou Medical University; Jingming Zhai, MD, Study Director — The First Affiliated Hospital of Henan University of Science and Technology
Locations (4):
- China (4):
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo Z, Shi Y, Song Z, Jia W, Wang S, Zhang Y, Ji X, Liu K, Zhang T, Cheng X, Zhao R. Single-incision robotic assisted surgery: a nonrandomized cohort pilot study on a novel surgical platform in colorectal surgery. Int J Surg. 2023 Nov 1;109(11):3417-3429. doi: 10.1097/JS9.0000000000000612. PMID 37526117